CLINICAL TRIAL: NCT05461040
Title: Optic Capture Without Anterior Vitrectomy in Pediatric Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ali Devebacak, Principal Investigator, Consultant Ophthalmologist, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OC3506
Record Dates: First submitted 2022-07-11; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Cataract, Juvenile
Keywords: cataract surgery; intraocular lens; optic capture; pediatric cataract; posterior capsulotomy
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optic capture of Intraocular lens without anterior vitrectomy (Group 1) (Experimental)
  Interventions: Procedure: optic capture
- in-the-bag implantation of Intraocular lens with anterior vitrectomy (Group 2). (Experimental)
  Interventions: Procedure: In-the-bag implantation of Intraocular lens

INTERVENTIONS:
Procedure: optic capture — optic capture of Intraocular lens without anterior vitrectomy
  Arms: Optic capture of Intraocular lens without anterior vitrectomy (Group 1)
Procedure: In-the-bag implantation of Intraocular lens — in-the-bag implantation of Intraocular lens with anterior vitrectomy
  Arms: in-the-bag implantation of Intraocular lens with anterior vitrectomy (Group 2).

SUMMARY:
Purpose: To compare two pediatric cataract surgery procedures: intraocular lens (IOL) optic capture without anterior vitrectomy (AV) and in-the-bag IOL implantation with AV.

Setting: Ege University Medical School Hospital, Izmir, Turkey. Design: Prospective randomized control clinical trial. Methods: Patients were randomly assigned to two groups: optic capture without AV (Group 1) or in-the-bag implantation with AV (Group 2). The following variables were compared: visual acuity, intraocular pressure, refractive errors, IOL tilt and decentration, lenticular astigmatism, anterior-posterior synechia, inflammatory cell deposits on IOL and post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital or developmental cataracts who had cataract surgery and primary IOL implantation at a tertiary care referral institute were included.

Exclusion Criteria:

* Traumatic or uveitic cataract, corneal opacity, iris coloboma, microphthalmia, microcornea, persistent fetal vascularization, congenital glaucoma, and retinopathy of prematurity were all considered exclusion criteria.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The prevalence of visual axis opacification | through study completion, an average of 2 years
  Eyes were evaluated for presence of visual axis opacification at the slit lamp examinations.
The prevalence of inflammatory deposits on Intraocular lens surface | through study completion, an average of 2 years
  Eyes were evaluated presence of inflammatory deposits between the margins of capsulorhexis at the slit lamp examinations.
The prevalence of anterior-posterior synechia | through study completion, an average of 2 years
  Eyes were evaluated for presence of anterior-posterior synechia at the slit lamp examinations.
Measurements of Intraocular lens tilt and decentration. | at the postoperative one-year
  Measurement of Intraocular lens (IOL) position at vertical and horizontal meridians at the Scheimpflug images captured with corneal topography. Scheimpflug images were obtained (Pentacam HR, Oculus Optikgerate Gmbh, Wetzlar, Germany) at one postoperative year. The horizontal and vertical meridians' photographs were analyzed.These images were processed in AutoCAD LT 2020 2D CAD software for IOL position assessment.(1) IOL Center: Two arches were drawn that fit perfectly on the anterior and posterior surfaces of the IOL. The points where these two arcs met were marked. Between these intersection points, a line was drawn. The midpoint of this line was accepted as the IOL center. (2) IOL Decentration: It was determined by measuring the distance (mm) from the IOL center point to the pupillary axis. (3) IOL Tilt: Angle (degree) between the IOL axis and the line passing through the iridocorneal angle.
Prediction error | at the post-operative one-month
  Refraction prediction error (PE) was found by subtracting the early post-operative refraction from the pre-operative target refraction.

SECONDARY OUTCOMES:
Intraocular pressure | at the postoperative one year
  Intraocular pressure was measured by Tonopen (Reichart Technologies, Depew, NY), Perkins handheld Mk2 tonometry (Haag-Streit, Koeniz, Switzerland) or Goldmann applanation tonometry (Haag Streit, Koeniz, Switzerland), considering the patient's age and compliance.
Lenticular astigmatism | One-year postoperatively
  Calculated by subtracting corneal astigmatism from manifest astigmatism.
Posterior segment complications | through study completion, an average of 2 years
  In the fundoscopic examination, the patients were evaluated for possible posterior segment complications such as retinal detachment, cystoid macular edema, and intraocular hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Devebacak, M.D., Principal Investigator — Ege University, Department of Ophthalmology
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided